CLINICAL TRIAL: NCT07263009
Title: Impact of Reflux Flow Volume on Semen Parameters Pre and Post Varicocelectomy
Brief Title: Reflux Flow Volume Impact on Semen Parameters Pre and Post Varicocelectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Adel Ragab Mohamed, Resident doctor, Assiut University
Other Study IDs: Scrotal duplex in varicocele
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Varicocele
Keywords: Scrotal duplex; Varicocele; Semen parameters; Reflux flow volume
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with bilateral clinical varicocele confirmed with scrotal color Doppler Ultrasonography

SUMMARY:
Evaluation of the impact of reflux flow volume and other ultrasonographic diagnostic parameters of varicocele on semen parameters before and 3 months varicocelectomy

DETAILED DESCRIPTION:
Varicocele is an abnormal dilatation and tortuosity of the pampiniform plexus of veins draining the testicles. It affects almost 15% of men in the general population, but its prevalence rises significantly reaching 35-40% among men with primary infertility and up to 80% of men with secondary infertility. Varicocele is known to have a deleterious effect on spermatogenesis through multiple mechanisms, resulting in a progressive decline in semen parameters. However, the precise pathophysiological impact of varicocele on male infertility is still unclear. Although clinical examination is considered the standard diagnostic method , a considerable number of varicocele can be detected via ultrasound. Color Doppler Ultrasonography (CDUS) is widely used as a non-invasive diagnostic tool for varicocele, mainly through detection of venous reflux which is a key diagnostic criterion. As the current CDUS-based grading systems rely on subjective and individual parameters which may not fully represent the harmful effect caused by the condition, there is a critical need for a more integrated and quantifiable parameter that can better predict the severity of testicular dysfunction and guide its treatment. Reflux flow volume is a quantitative parameter measured via the CDUS, referring to the rate of retrograde blood flow passing through the dilated veins during reflux episodes. This parameter integrates reflux duration, velocity and vein diameter. Thus, it can provide a more comprehensive assessment of reflux severity than any of the individual components alone. Consequently, reflux flow volume can serve as a reliable marker for testicular function. By investigating its relation to other ultrasonographic parameters, testicular volume and their impact on semen parameters, testosterone and follicle stimulating hormone (FSH) levels, it has the potential to transform diagnostic strategies and predict the impact of varicocelectomy on spermatogenesis and hormonal changes. Therefore, it can stratify patients for the therapeutic approach and provide a better prognostic tool for varicocele management

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral clinical varicocele confirmed by Scrotal Color Doppler Ultrasonography

Exclusion Criteria:

* Unilateral varicocele.
* Recurrent varicocele.
* History of undescended testis, orchitis, testicular trauma, torsion or scrotal surgery.
* Inguinal hernia, hydrocele or scrotal mass.
* Prior chemotherapy, radiotherapy or any other gonadotoxic agents.
* Uncontrolled systemic illness.
* Chromosomal or genetic anomalies.
* Azoospermia and severe oligozoospermia (< 5 million/ml)

Ages: 20 Years to 50 Years | Sex: Male
Age Groups: Adult
Study Population: Male patients with bilateral clinical varicocele confirmed with scrotal color doppler Ultrasonography
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Scrotal ultrasonographic parameter | Preoperative
  Reflux volume(ml/min)

SECONDARY OUTCOMES:
Semen parameter | Preoperative and 3 months postoperative
  Sperm concentration (million/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Adel, Principal Investigator — Assiut University

REFERENCES:
- [Background] Senturk AB, Cakiroglu B, Yaytokgil M, Aydin C, Sungur M, Akkoc A. Effect of venous reflux time on testosterone and semen parameters of infertile males after microscopic varicocelectomy. Andrologia. 2020 Jul;52(6):e13583. doi: 10.1111/and.13583. Epub 2020 Apr 9. PMID 32271466
- [Background] Bagheri SM, Khajehasani F, Iraji H, Fatemi I. A Novel Method for Investigating the Role of Reflux Pattern in Color Doppler Ultrasound for Grading of Varicocele. Sci Rep. 2018 Apr 25;8(1):6517. doi: 10.1038/s41598-018-24890-2. PMID 29695731
- [Background] Kocakoc E, Serhatlioglu S, Kiris A, Bozgeyik Z, Ozdemir H, Bodakci MN. Color Doppler sonographic evaluation of inter-relations between diameter, reflux and flow volume of testicular veins in varicocele. Eur J Radiol. 2003 Sep;47(3):251-6. doi: 10.1016/s0720-048x(02)00182-1. PMID 12927671